CLINICAL TRIAL: NCT02938325
Title: Monitoring Awareness and Pain Under Anesthesia Using a New EEG Based System
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Rambam Health Care Campus (Other)
Responsible Party: Sponsor
Other Study IDs: 152-16 rambam-CTIL
Record Dates: First submitted 2016-09-26; First posted 2016-10-19 (Estimated); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Awareness Under Anesthesia
Keywords: Electroencephalogram; awareness

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- No intervention: General Anesthesia: Thirty patients undergoing elective surgery under general anesthesia who will be monitored with standard ASA, BIS and EEG for comparisons. In recovery unit, at the end of the surgery, patients will be questioned for awareness under anesthesia by Modified Brice Questionnaire.
  There will be no intervention. Patients will be anesthetized with general anesthesia as they were supposed to be for their elective surgery. The EEG during the anesthesia will be assessed afterwards, and patients will be asked about their memory from the surgery.
- No intervention: Sedation: Fourty patients undergoing elective cardiac catheterization under conscious sedation who will be monitored with standard ASA, BIS and EEG for comparisons. In recovery unit, at the end of the procedure, patients will be questioned for awareness under sedation by Modified Brice Questionnaire.
  There will be no intervention. Patients will be anesthetized with sedation as they were supposed to be for their elective cardiac catheterization. The EEG during the anesthesia will be assessed afterwards, and patients will be asked about their memory from the surgery.
- No Intervention - Awake Volunteers: EEG and BIS will be recorded in twenty volunteers, for 10 minutes, in supine position, while their eyes are closed. This recording will be utilized as for positive control for recall.

SUMMARY:
General anesthesia (GA) is the process of induction of unconsciousness in order to undergo surgery. Unlike sleep, a process of "anesthesia" is not related at all, 'Sleep' and does not include dreams - but is done by using drugs that cause a kind of "unconsciousness" control.

The induction of GA includes combination of drugs - for sleep (inhalation anesthesia or hypnotic drugs intravenously), analgesia (opiates) and muscle relaxants. Since most of our patients paralyzed during surgery, the anesthesiologists have no way of knowing whether our paralyzed patient is asleep or awake. If the patient is awake and paralyzed, a situation named "awareness under anesthesia" it can cause him a traumatic experience that would leave him a cripple for his whole life.

There are many stories about patients who lay paralyzed, awake, while been operated, who remembered every word of what happened during the operation and of course could not mark the anesthetist that they are awake. The anesthesiologist might suspect that his patient is awake and paralyzed through "signals" from the sympathetic nervous system - for example the increase in heart rate and blood pressure. But many of our patients receive different medications (eg, beta-receptor blockers that does not allow the rise of a pulse) obscuring the clinical signs, so that the patient is awake and paralyzed without being noticed by the anesthesiologist.

Some patients are at a higher risk to suffer from awareness under anesthesia, because the anesthesiologist cannot provide "enough" anesthesia, due to their medical condition, for example: women in caesarean section under GA, patients in cardiac surgery or injured trauma patients.

Twenty years ago, an EEG based tool, naming "BIS" was developed. Nowadays, BIS monitor's credibility is questionable 1. The effect of different hypnotic drugs is not uniform. 2. Recently it was shown that a paralyzed patient BIS index could fall mimicking a situation of a sleep - enabling a paralyzed patient being awake. Thus, it is not clear whether the calculation of the BIS monitor is based on physiological models that define what is consciousness, loss of consciousness and how consciousness arises. It seems that the BIS is only suitable for certain drugs - not as a general monitor for the level of anesthesia.

The purpose of the present study is to develop a universal system for determining awareness under GA using an innovative algorithm for analyzing EEG waves, based on the physiological processes of attention and perception underlying the basis for sedation and GA.

ELIGIBILITY:
Inclusion Criteria:

* ASA 1-3
* Patients for elective surgery under general anesthesia or elective procedures under sedation (such as cardiac electrical studies, liver chemo-embiolization, biliary tract drainage)
* The willing of the patient to fulfil the Modified Brice Questionnaire at the end of the procedure in recovery unit
* Healthy volunteers that will accept to be monitored with EEG and BIS for 10 minutes in supine position, as control.

Exclusion Criteria:

* Lack of consent
* Emergent surgery Emergent procedure (catheterization)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients undergoing elective procedures under sedation, or patients undergoing surgery under general anesthesia. Another twenty volunteers will undergo elective EEG and BIS recording for 10 minutes, for comparison.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Could a new EEG based Posteriorization/Anteriorization (P/A) index identify recall under sedation | Immediately after surgery
  Posteriorization/ Anteriorizatio index is analyzed at the end of the surgery, with no influence on the intraoperative treatment of the patient.

SECONDARY OUTCOMES:
The association between the P/A index to muscle activity | Sub- analysis, within 6 months from the date the last patient was recruited for the study
  The correlation between the electromyelograph (EMG) activity, to the calculated index
The association between BIS to muscle activity | Sub- analysis, within 6 months from the date the last patient was recruited for the study
  The correlation between the electromyelograph (EMG) activity, to BIS
Could Bis identify recall under sedation | Immediately after surgery
  BIS index is recorded during the procedure, but the anesthesiologists is blinded to its results. The association between BIS and recall is analyzed at the end of the surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Dana Baron Shahaf, MD PhD, Principal Investigator — Rambam Health Care Campus
Locations (1):
- Rambam Health Care Campus, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] White NS, Alkire MT. Impaired thalamocortical connectivity in humans during general-anesthetic-induced unconsciousness. Neuroimage. 2003 Jun;19(2 Pt 1):402-11. doi: 10.1016/s1053-8119(03)00103-4. PMID 12814589
- [Background] Alkire MT, Hudetz AG, Tononi G. Consciousness and anesthesia. Science. 2008 Nov 7;322(5903):876-80. doi: 10.1126/science.1149213. PMID 18988836
- [Background] Shalbaf R, Behnam H, Jelveh Moghadam H. Monitoring depth of anesthesia using combination of EEG measure and hemodynamic variables. Cogn Neurodyn. 2015 Feb;9(1):41-51. doi: 10.1007/s11571-014-9295-z. Epub 2014 May 9. PMID 26052361
- [Background] Osterman JE, Hopper J, Heran WJ, Keane TM, van der Kolk BA. Awareness under anesthesia and the development of posttraumatic stress disorder. Gen Hosp Psychiatry. 2001 Jul-Aug;23(4):198-204. doi: 10.1016/s0163-8343(01)00142-6. PMID 11543846
- [Background] Avidan MS, Palanca BJ, Glick D, Jacobsohn E, Villafranca A, O'Connor M, Mashour GA; BAG-RECALL Study Group. Protocol for the BAG-RECALL clinical trial: a prospective, multi-center, randomized, controlled trial to determine whether a bispectral index-guided protocol is superior to an anesthesia gas-guided protocol in reducing intraoperative awareness with explicit recall in high risk surgical patients. BMC Anesthesiol. 2009 Nov 30;9:8. doi: 10.1186/1471-2253-9-8. PMID 19948045
- [Background] Newton DE, Thornton C, Konieczko K, Frith CD, Dore CJ, Webster NR, Luff NP. Levels of consciousness in volunteers breathing sub-MAC concentrations of isoflurane. Br J Anaesth. 1990 Nov;65(5):609-15. doi: 10.1093/bja/65.5.609. PMID 2248835
- [Background] Dupont H. [Anesthesia awareness and the bispectral index]. Ann Fr Anesth Reanim. 2008 Dec;27(12):1042-3. doi: 10.1016/j.annfar.2008.10.013. No abstract available. French. PMID 19097272
- [Background] Short TG, Campbell D, Leslie K. Response of bispectral index to neuromuscular block in awake volunteers. Br J Anaesth. 2016 May;116(5):725-6. doi: 10.1093/bja/aew089. No abstract available. PMID 27106988
- [Background] Suzuki M, Edmonds HL Jr, Tsueda K, Malkani AL, Roberts CS. Effect of ketamine on bispectral index and levels of sedation. J Clin Monit Comput. 1998 Jul;14(5):373. doi: 10.1023/a:1009975701184. No abstract available. PMID 9951765
- [Background] Voss L, Sleigh J. Monitoring consciousness: the current status of EEG-based depth of anaesthesia monitors. Best Pract Res Clin Anaesthesiol. 2007 Sep;21(3):313-25. doi: 10.1016/j.bpa.2007.04.003. PMID 17900011
- [Background] Chen Y, Cai A, Dexter F, Pryor KO, Jacobsohn EM, Glick DB, Willingham MD, Escallier K, Winter A, Avidan MS. Amnesia of the Operating Room in the B-Unaware and BAG-RECALL Clinical Trials. Anesth Analg. 2016 Apr;122(4):1158-68. doi: 10.1213/ANE.0000000000001175. PMID 26859877
- [Background] Brunner M, Vaughan D. Evoked potential monitoring in anaesthesia and analgesia. Anaesthesia. 2000 Aug;55(8):823-5. doi: 10.1046/j.1365-2044.2000.01629-27.x. No abstract available. PMID 10947725
- [Background] Shahaf G, Pratt H. Thorough specification of the neurophysiologic processes underlying behavior and of their manifestation in EEG - demonstration with the go/no-go task. Front Hum Neurosci. 2013 Jun 24;7:305. doi: 10.3389/fnhum.2013.00305. eCollection 2013. PMID 23805094
- [Background] Shahaf G, Fisher T, Aharon-Peretz J, Pratt H. Comprehensive analysis suggests simple processes underlying EEG/ERP - demonstration with the go/no-go paradigm in ADHD. J Neurosci Methods. 2015 Jan 15;239:183-93. doi: 10.1016/j.jneumeth.2014.10.016. Epub 2014 Nov 1. PMID 25445244